CLINICAL TRIAL: NCT05019274
Title: The Impact of Culinary Medicine vs. Nutrition Education on Diabetes Outcomes: A Randomized Trial
Brief Title: Culinary Medicine vs. Nutrition Education in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Michael Edward Bowen, Assistant Professor Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU-2020-1244
Record Dates: First submitted 2021-07-30; First posted 2021-08-24 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Primary Disease: 1. Type 2 Diabetes
Keywords: Type 2 diabetes; culinary medicine; medical nutrition therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This pragmatic effectiveness trial randomizes patients 1:1 to a series of 6 virtual Culinary Medicine classes or 6 standard of care nutrition visits .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culinary Medicine (Experimental): Series of 6 virtual group Culinary Medicine sessions delivered monthly for 6 months
  Interventions: Other: Culinary Medicine Intervention
- Nutrition Education (Active Comparator): Series of 6 standard of care nutrition visits delivered by clinic dieticians. These are a mix of individual and group sessions.
  Interventions: Other: Standard of Care Nutrition Visits

INTERVENTIONS:
Other: Culinary Medicine Intervention — Participants randomized to the Culinary Medicine intervention will complete a series of 6 virtual culinary medicine cooking classes (1 class per month for 6 months). Virtual sessions will be delivered via Zoom using a combination of large group instruction and small group break-out sessions in which participants prepare a recipe in their home kitchen with the virtual assistance from trained group facilitators. After preparing the dish, participants will enjoy the dish they prepared and report-back to the large group about their dish and experience. Classes will be conducted in English and Spanish with language-concordant instructors and facilitators.
  Arms: Culinary Medicine
Other: Standard of Care Nutrition Visits — Participants randomized to standard of care nutrition visits will complete a series of 6 nutrition visits (1 session per month for 6 months) led by bilingual (English/Spanish) dieticians. Sessions will consist of a mix of individual and small group sessions per standard of care in the clinic.
  Arms: Nutrition Education

SUMMARY:
This pragmatic trial compares the effectiveness of virtual culinary medicine classes vs. standard of care medical nutrition visits to improve glycemic control in patients with uncontrolled type 2 diabetes . Culinary medicine teaches healthy eating principles through a combination of experiential cooking classes and focused didactic sessions. The primary study outcome is glycemic improvement (A1c). Qualitative evaluation will assess participant experience, impact, and durability of behavior changes related to nutrition. A short term cost analysis will be conducted to inform program costs and cost effectiveness.

DETAILED DESCRIPTION:
A total of 130 participants with uncontrolled type 2 diabetes will be recruited from a safety-net health system that provides comprehensive care for the uninsured and underinsured residents of Dallas County, Texas. Eligible participants will be actively engaged in primary care and recruited from clinical practice. Participants will be randomized to two arms: Culinary Medicine and standard of care medical nutrition therapy (MNT). Certified culinary medicine instructors will deliver a series of 6 monthly Culinary Medicine classes virtually with participants cooking in their own homes. A series of 6 standard of care medical nutrition sessions will be delivered by the health system using a combination of individual and group sessions both in person and virtually. All participants will be enrolled in a 12 month food assistance program in partnership with community based partners to provide access to healthy foods. Classes will be delivered over 6 months, and participants will be followed for an additional 6 months to assess the durability of glycemic response and behavior changes. A cost analysis will examine the system cost to deliver the intervention and the short term cost effectiveness examining the cost per participant achieving a clinically meaningful reduction in A1c.

ELIGIBILITY:
Inclusion Criteria:

* No nutrition visit in the past 12 months.
* Hemoglobin A1C ≥ 7.5% within the past six months.
* Diagnosed with established Type 2 Diabetes > 12 months
* Receiving primary care at Hatcher Station Health Center and an assigned primary care provider within the past 18 months.
* Completion of at least 2 of the 4 Health Living with Diabetes (HLWD) virtual and/or in-person sessions.

Exclusion Criteria:

* Patients who cannot hear virtual and/or in-person instruction
* Patients who cannot read or speak English or Spanish
* Patients who are unable to understand study information
* Patients younger than 18 years of age
* Patients who are unable to communicate with voice (for participation in phone surveys, focus groups and semi-structured interviews)
* Patients without access to a smart phone or other device with internet and/or data capability to participate in virtual classes
* We will exclude patients with chronic kidney disease (CKD) stage 4 or 5 (eGFR < 30 or on dialysis) because their renal function may require additional nutritional counseling and dietary modifications beyond the scope of the proposed culinary medicine and nutrition sessions delivered in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 3, 6, and 12 months
  A1c will be measured at baseline, 3, 6 and 12 months. Change in A1c will be assessed at 6 months (end of active intervention) and also at 12 months (i.e. 6 months after completion of active intervention) to assess the durability of the intervention on glycemic control. Pre-specified subgroup analyses will also examine A1c outcomes by: 1) prior participation in diabetes education and nutrition education. Stratified analyses by number of sessions attended will also be conducted.

SECONDARY OUTCOMES:
Change in weight | 3, 6, and 12 months
Change in BMI | baseline, 6 and 12 months
Change in blood pressure | baseline, 6, and 12 months
Food security score | baseline, 6 months and 12 months
  U.S. Household Food Security Survey Module: Six-Item Short Form. The score ranges from 0 to 6 with 0 indicating high food security and 6 indicating very low food security.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Bowen, MD, Principal Investigator — UT Southwestern Medical Center in Dallas
Locations (1):
- Parkland Health and Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No